CLINICAL TRIAL: NCT02441842
Title: Evaluation of Perioperative Biochemical Stress Factors in Craniotomy Neurosurgical Procedure With Respect to Preoperative Hypertension
Brief Title: Evaluation of Periop Biochemical Stress Factors in Craniotomy Neurosurgical Procedure With Respect to Preop Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sanjib Adhikary, Assist Prof; Dir. Acute Pain, Regional Anesthesia/ Orthopedics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5820 / 2006
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Perioperative Hypertension
Keywords: β-blocker; ACE inhibitor; Stress; Craniotomy; Postop hypertension; neurosurgical patients
MeSH Terms: interventions — Atenolol; Lisinopril; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A : Atenolol (Active Comparator): oral atenolol (50mg)
  Interventions: Drug: atenolol
- Group C: Placebo (Placebo Comparator): glucose tablet (10mg)
  Interventions: Other: glucose
- Group L: Lisinopril (Active Comparator): oral lisinopril (5mg)
  Interventions: Drug: lisinopril

INTERVENTIONS:
Drug: atenolol — administered 60 minutes pre procedure
  Arms: Group A : Atenolol
Drug: lisinopril — administered 60 minutes pre procedure
  Arms: Group L: Lisinopril
Other: glucose — administered 60 minutes pre procedure
  Arms: Group C: Placebo

SUMMARY:
Perioperative hypertension is commonly associated with surgical craniotomy. As the sympathetic nervous system and the renin-angiotensin-aldosterone system play a key role in the development of this hypertension, preoperative single dose therapy with a -adrenergic receptor blocker or an angiotensin converting enzyme (ACE) inhibitor may be useful in preventing this. To assess this as well as to study potential markers of these two systems, the investigators will perform a randomized, double blind, placebo controlled study to compare the single dose effect of preoperative administration of a -receptor blocking drug (atenolol) and an ACE inhibitor (lisinopril) with a control group receiving a placebo tablet (glucose) on perioperative hypertension in craniotomy patients.

DETAILED DESCRIPTION:
All patients included in the study will be visited 12 hours preoperatively for determination of base-line (preoperative) blood pressure and heart rate, at which time a blood sample will be taken and the patients will be randomized. The next day, sixty minutes prior to surgery, all patients will receive oral diazepam (10mg) and the blinded study medication. This medication was previously prepared by an independent pharmacist, and dispensed in appropriate packaging. Thus, Group C, the control group, will receive a glucose tablet (10mg), Group A, will receive oral atenolol (50mg) and Group L will receive oral lisinopril (5mg). An intravenous cannula will be placed and normal saline will be infused at the rate of 60 - 70 ml/hr. Haemodynamics (blood pressure and heart rate) will be monitored using a multichannel monitor (and the patient's radial artery (non-dominant arm) will be cannulated for further blood sampling and blood pressure monitoring (Agilent Technologies, MA, USA). Anaesthesia will beinduced with thiopental (4-5 mg.kg-1) and fentanyl, (1-2μg.kg-1). Vecuronium, (0.06-0.1 mgkg-1) will be administered to facilitate tracheal intubation and to maintain neuromuscular blockade. Isoflurane (0.7 - 1.2 MAC) will be administered to maintain the Bispectral Index (BIS) (Aspect Medical System Inc, MA, USA), within the range of 35 - 45. End tidal CO2 partial pressure will be maintained between 4-4.6 kPa (IntelliVue Anesthetic Gas Modules-G1, Redmond, WA, USA). During the surgery, intravenous fentanyl and vecuronium will be administered at the discretion of the anaesthetist for pain control and muscle relaxation respectively. An increase in mean arterial pressure (MAP) in excess of 20% of the pre-operative value will be treated either by increasing the inspired isoflurane concentration or by administering metoprolol. Additionally, a decrease in MAP exceeding 20% will be treated by reducing the isoflurane inspired concentration or by the administration of ephedrine in small doses (2.5-4mg). Ondansetron (4mg) will be administered 45 minutes before the expected conclusion of surgery and neuromuscular agents will be reversed using 2.5 mg of neostigmine and 0.4 mg of glycopyrrolate at the end of skin suturing. Isoflurane will be discontinued at the last suture, and patients will be extubated when they respond to verbal stimulation or coughed. The total amount and type of fluids administered during the procedure will be recorded.

The MAP, HR, end-tidal isoflurane, and end tidal CO2 will be recorded every 10 min following induction until extubation, and MAP and HR only, every 30 min after admission to the neuro-intensive care unit for 12 hrs. These data will be collected from the monitors using printouts after each case and the anesthesia record will also be photocopied. Postoperative pain will be treated with paracetamol (1gm) administered rectally every 6 hrs and morphine injection (2.5mg) intravenously as required.

Hypertension is defined as any mean arterial blood pressure (MAP) more than 20% of the preoperative value (determined 12hrs before the surgery, vide supra).

Blood samples (3 ml) will be collected from each patient pre operatively from venapuncture (12hrs before the surgery), and intra-operatively at the time of dural opening, and immediately after extubation, via the arterial line. Collected blood samples will immediately be centrifuged and stored at -70°C for analysis of plasma renin, aldosterone, norepinephrine, and serum sodium concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo craniotomy for a supratentorial brain tumor resection
* Weight between the limits of 70 - 100 kgs

Exclusion Criteria:

* Weight less than 70 kgs or more thank 100 kgs
* Meds for hypertension
* Evidence of raised intracranial pressure, hypertension, cardiovascular, endocrine or renal disease

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
MAP changes | time of incision, extubation and 12 hours postop
  MAP changes associated with preoperative single dosage treatment with atenolol or lisinopril, at the time of dural incision and at extubation, as well as 12 hours postoperatively compared to the control group
HR changes | time of incision, extubation and 12 hours postop
  HR changes associated with preoperative single dosage treatment

SECONDARY OUTCOMES:
plasma concentrations of vasoactive markers | 12 hours before procedure, during time of dural opening and immediately following extubation
  blood sample taken
plasma concentrations of serum sodium levels | 12 hours before procedure, during time of dural opening and immediately following extubation
  blood sample taken

CONTACTS AND LOCATIONS:
Overall Officials: K.V. Parthiban, PhD, Principal Investigator — Christian Medical College, Dept of Neurological Sciences